CLINICAL TRIAL: NCT00076531
Title: Clinical Trial for Prostate Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Oakwood Laboratories, LLC (Industry)
Masking: None | Purpose: Treatment
Other Study IDs: OL-007
Record Dates: First submitted 2004-01-26; First posted 2004-01-27 (Estimated); Last update posted 2008-01-28 (Estimated); Status verified 2008-01

CONDITIONS: Prostate Cancer
Keywords: Prostate; Cancer; PSA; Leuprolide
MeSH Terms: conditions — Prostatic Neoplasms; Neoplasms | interventions — Leuprolide

INTERVENTIONS:
Drug: Leuprolide Acetate for Injectable Suspension 22.5 mg

SUMMARY:
Phase III trial using an injectable for treatment of prostate cancer.

Min Age: 40 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2003-12; Primary Completion 2004-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James A. Page, M.D., Study Chair — Oakwood Laboratories, LLC

REFERENCES:
- See also: Oakwood (sponsor) site — http://www.oakwoodlabs.com